CLINICAL TRIAL: NCT03194360
Title: Risk Factors of Delirium in Sequential Sedation Patients in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Kang Yan, Study Chair: Y Kang, Dr Critical Medicine Department,West China Hospital of Sichuan University, West China Hospital
Other Study IDs: HuaxiICM
Record Dates: First submitted 2017-06-17; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Delirium; Mechanical Ventilation; Sedation
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- delirium group
- nondelirium group

SUMMARY:
Delirium is one of main adverse events in ventilated patients who receive long-term usage of mono-sedative. Sequential sedation may reduce these adverse effects. This study aimed to evaluate incidence and risk factors for delirium in sequential sedation patients.

DETAILED DESCRIPTION:
Previous studies have showed that patients under mechanical ventilation have a higher risk for experiencing delirium than nonmechanically ventilated patients (20%-50%). Its occurrence is also more frequent in elder patients. More than that, it is often hard to identify delirium by physicians, leading to unreasonable management of ICU patients.

And delirium is one of main adverse events in ventilated patients who receive long-term usage of mono-sedative. Sequential sedation may reduce these adverse effects.

However, few present studies focus on delirium in sequential sedation patients. Thus, in this study, we aimed to determine the factors of delirium in patients who received sequential sedation in ICU.

ELIGIBILITY:
Inclusion Criteria:

1. Intubated patients;
2. Age≥18 years old;
3. Anticipated Ventilation and sedation duration of at least 72 hours.

Exclusion Criteria:

1. Allergy to the study drug;
2. suspected pregnancy;
3. gross obesity;
4. Extremely unstable of circulatory system, such as systolic blood pressure less than 90 mm Hg despite plasma volume expansion and continuous infusions of vasopressors before the start of study drug infusion;
5. Uncontrolled abnormal hypertension, such as systolic blood pressure more than 180 mmHg or diastolic more than105 mmHg;
6. Heart rate less than 50 bpm;
7. Second or third degree heart block;
8. moribund state;
9. history of alcoholism or intake of anti-anxiety drugs or hypnotics;
10. chronic renal failure;
11. coma by cranial trauma or neurosurgery or unknown etiology or epileptic state;
12. History of neuromuscular disease;
13. unwillingness to provide informed consent by patients or their authorized surrogates following ICU admission.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with an age greater than 18 years old and less than 80 years old, who were expected to receive mechanical ventilation longer than 72 hours and accepted sedation therapy were recruited on admission to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Delirium assessment in Sequential Sedation Patients | A maximum of twenty-eight days or until ICU discharge, whichever occurred first.
  The primary outcome of this study was delirium. Patient evaluations were implemented using Confusion Assessment Method for the Intensive Care Unit (CAM-ICU) scale every four hours a day for a maximum of twenty-eight days or until ICU discharge, whichever occurred first. The risk factors were analyzed using risk regression (logistic-regression). Any variables which had P<0.2 after univariable logistic-regression or potential variables associated with delirium were included for multivariable logistic-regression. P<0.05 was considered to represent statistical significance.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Critical care medicine of West China Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou Y, Jin X, Kang Y, Liang G, Liu T, Deng N. Midazolam and propofol used alone or sequentially for long-term sedation in critically ill, mechanically ventilated patients: a prospective, randomized study. Crit Care. 2014 Jun 16;18(3):R122. doi: 10.1186/cc13922. PMID 24935517
- [Result] Mehta S, Cook D, Devlin JW, Skrobik Y, Meade M, Fergusson D, Herridge M, Steinberg M, Granton J, Ferguson N, Tanios M, Dodek P, Fowler R, Burns K, Jacka M, Olafson K, Mallick R, Reynolds S, Keenan S, Burry L; SLEAP Investigators; Canadian Critical Care Trials Group. Prevalence, risk factors, and outcomes of delirium in mechanically ventilated adults. Crit Care Med. 2015 Mar;43(3):557-66. doi: 10.1097/CCM.0000000000000727. PMID 25493968
- [Result] Ely EW, Gautam S, Margolin R, Francis J, May L, Speroff T, Truman B, Dittus R, Bernard R, Inouye SK. The impact of delirium in the intensive care unit on hospital length of stay. Intensive Care Med. 2001 Dec;27(12):1892-900. doi: 10.1007/s00134-001-1132-2. Epub 2001 Nov 8. PMID 11797025
- [Result] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966